CLINICAL TRIAL: NCT06943989
Title: Pulmonary and Inflammatory Responses Following Exposure to a Low Concentration of Ozone or Clean Air for 6.6 Hours at Rest in Healthy Young Adults.
Brief Title: Pulmonary and Inflammatory Responses Following Exposure to a Low Concentration of Ozone or Clean Air at Rest
Acronym: LOCONOZ3
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jairus Pulczinski, Research Biologist, Environmental Protection Agency (EPA)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: EnvironmentalPA
Record Dates: First submitted 2025-04-17; First posted 2025-04-25 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Lung Inflammation; Experimental Lung Inflammation
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.070 ppm ozone concentration (Experimental): Exposure to 0.070 ppm ozone for 6.6 hours at rest
  Interventions: Other: Ozone Exposure
- Clean air (0.0 ppm ozone) (Experimental): Exposure to clean air (0.0 ppm ozone) for 6.6 hours while at rest
  Interventions: Other: Clean air (0.0 ppm ozone)

INTERVENTIONS:
Other: Ozone Exposure — 6.6 hour exposure to 0.07 ppm ozone while at rest
  Arms: 0.070 ppm ozone concentration
Other: Clean air (0.0 ppm ozone) — 6.6 hour exposure to clean air (0.00 ppm ozone) while at rest
  Arms: Clean air (0.0 ppm ozone)

SUMMARY:
The primary purpose of this study is to measure pulmonary function, symptoms, and pulmonary inflammatory responses in healthy young adults during and immediately after exposure to a low concentration of ozone (0.070 ppm) or clean air for 6.6 hours while at rest. This concentration is the current EPA NAAQS standard for ozone.

DETAILED DESCRIPTION:
Potential health effects of ozone have been extensively studied over decades at various levels of exposure concentration for varying time periods while at varying levels of exertion. The effects of ground level ozone exposure have been well documented, particularly for decrements in lung function and for markers of pulmonary inflammation, such as neutrophils in sputum. (1) The majority of previous studies were done at ozone concentrations between 0.12 and 0.40 ppm, for one to four hours of exposure, with moderate to intermittent exercise to simulate daily activities. These concentrations are considerably higher than the level of the current EPA National Ambient Air Quality Standards (NAAQS) ozone standard of 0.07 ppm (8-hour average). Only a small number of studies have assessed changes in lung function and inflammatory markers following longer exposure to ozone (2-10). These latter studies have shown that exposure to low concentrations of ozone for 6.6 hours at concentrations between 0.06 and 0.08 ppm while performing moderate exercise causes mild reversible decrements in lung function (<5%) as measured by forced vital capacity (FVC) and forced expired volume at 1 s (FEV1) assessed immediately after exposure in healthy young adults. There are also many studies of ozone exposures which included healthy adults at rest that report a mix of respiratory effects, but these studies were carried out at very high concentrations ranging from 0.1 to 1.0 ppm for one-to-two-hour durations ppm is the lowest concentration eliciting lung function decrements in controlled human exposure studies of one-to-two-hour exposure with participants at rest (not exercising). Taken together, the controlled human exposure evidence suggests that ozone-induced respiratory effects are determined by the ozone concentration as well as the exposure duration and activity level of exposed participants.

In the 2015 and 2020 O3 NAAQS reviews, the strongest evidence of respiratory effects causally related to short-term O3 exposures came from controlled human exposure studies reporting an array of respiratory effects in study participants while exercising moderately. The 2015 decision to revise the level of the standard to 70 ppb (and the 2020 decision to retain this standard), relied on 70 ppb being below the O3 exposure concentration (80 ppb) shown in 6.6 hour controlled human exposure studies with moderate exercise to result in the widest range of respiratory effects and below the lowest O 3 exposure concentration (73 ppb) shown to result in the adverse combination of lung function decrements and respiratory symptoms.

In 2021, the EPA Administrator decided to reconsider the 2020 decision to retain the current O3 NAAQS. As part of that process EPA released a draft Policy Assessment (PA) for the Reconsideration of the Ozone National Ambient Air Quality Standards v.2 (draft PA) that concluded that the available evidence was largely unchanged since the 2015 and 2020 reviews provided support for retaining the current primary standard. As part of the reconsideration process, EPA had provisionally considered a recent controlled human exposure study by Hernandez et al., (2021) which reported a small but significant change in lung function (FEV1 decrement) in 14 participants exposed largely at rest to an average O3 concentration of 70 ppb for 6.6 hours (Duffney Memo 2021). EPA noted that this study was designed to test the responsiveness of air quality sensors under rapidly changing air quality conditions and utilized an unusual exposure protocol that differed from protocols used in other controlled human exposure studies, including those with or without exercise.

Specifically, the O 3 concentrations were changed from 60 ppb to 80 ppb then back to 60 ppb during each hour of the study. This pattern and magnitude of varying concentrations are unlike patterns observed in ambient air, and it is unclear how this may have affected the observed responses.

The Clean Air Scientific Advisory Committee (CASAC) was established under the Clean Air Act Amendments of 1977 to provide independent advice to the EPA Administrator. The CASAC reviewed the 2021 draft PA on ozone and provided their advice in a June 2023 report. Relying in part on the Hernandez et al study (10), the CASAC recommended that the level of the current 0.07 ppb standard was not adequate to protect public health and that the NAAQS be revised. In particular, the CASAC noted that the small but significant decrement in FEV1 in participants exposed to an average 0.07 ppm O3 concentration for 6.6 hours while at rest (without exercise) called into question the assumption that moderate to heavy exercise is necessary for adverse health effects to occur at low levels of O3 exposure. The EPA is considering whether a level of 0.07 ppm provides adequate protection for public health. EPA researchers have been asked to conduct a study similar to those previously done at ozone exposure concentrations of 0.06, 0.07, and 0.08 ppm with healthy volunteers, but with volunteers at rest, rather than exercising. EPA believes such a study would provide clinical evidence for whether moderate to heavy exercise is necessary for adverse health effects to occur at the current level of the ozone standard.

ELIGIBILITY:
Inclusion criteria:

* Age 18-35 years old healthy male and female.
* No concerning findings on electrocardiogram (ECG) and no history of serious heart arrythmia.
* Normal lung function based on current American Thoracic Society(ATS) criteria.

  * Forced vital capacity (FVC) 80% of that predicted for age, gender and height.
  * Forced expiratory volume in one second (FEV1) 80% of that predicted for age, gender and height.
  * FEV1/FVC absolute ratio of at least 70%.
* Oxygen saturation normal (94%) at the time of physical exam.

Exclusion criteria:

* A history of acute or chronic cardiovascular disease, chronic respiratory disease, a history of hospitalization for COVID-19, diabetes, rheumatologic diseases, immunodeficiency state.
* Active asthma or a history of asthma within the past ten years (by spirometry, medication use
* and/or symptoms).
* Allergy to chemical vapors or gases.
* Currently pregnant, attempting to become pregnant or breastfeeding.
* The use of high doses of vitamins and supplements, homeopathic/naturopathic medicines or medications (e.g., steroids, beta blockers) which may impact the results of the ozone challenge or interfere with any other medications potentially used in the study.
* Medications not specifically mentioned here will be reviewed by the investigators prior to a participant's inclusion in the study.
* Active smoker or smoking within the previous 2 years, or participants with a lifetime smoking
* history equivalent to 10 pack-years or greater. This includes vaping, hookah use and e-cigarette use.
* Uncontrolled hypertension (= 140 systolic, = 90 diastolic). Blood pressure readings equal to or greater that 140 Systolic and equal to or greater that 90 diastolic.
* Inability to communicate verbally in English.
* Unspecified illnesses or chronic conditions which, in the judgment of the investigators and EPA clinical staff, might increase the risk associated with ozone inhalation or affect the study outcome measurements.
* Individuals who will NOT comply with the following temporary exclusion criteria:

Temporary exclusion criteria:

* Individuals who have had an acute respiratory illness within 4 weeks.
* Individuals who have active allergic rhinitis and/or conjunctivitis.
* Individuals unable to avoid drinking alcohol for 24 hours prior to all study visits.
* Individuals who have been exposed to smoke and fumes for 24 hours before all visits.
* Individuals who have used an ozone-based home air purifier for 24 hours before all visits.
* Individuals who have consumed any food in the 2 hours prior to the consenting visit and follow up visit (contraindicated for sputum induction).
* Individuals should refrain from all over the counter anti-inflammatory agents (e.g., ibuprofen, aspirin, naproxen, acetaminophen) and antihistamines for allergies (e.g., cetirizine, diphenhydramine), and antioxidants for a period of one week prior to the consenting visit and to the exposure visits.
* Individuals who have been exposed to or have consumed any agent or have undertaken any recent activity in advance of any study visit that the investigators believe may compromise participant safety and/or study results.
* Individuals with a total symptom score greater than or equal to 20, or with more than one score equal to 3, with the exception of the symptom score for sweating.
* Failure to arrive at the medical station within 15 minutes of their scheduled visit time.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
FVC | measured (pre) before starting 6.6 hours of exposure, , immediately after (post), and at follow up 24 hours later (Follow Up)
  forced vital capacity
FEV1 | measured (pre) before starting 6.6 hours of exposure, , immediately after (post), and at follow up 24 hours later (Follow Up)
  forced expiratory volume in 1 second

SECONDARY OUTCOMES:
% neutrophils collected by induced sputum | 18 hours post exposure
  Subjects will breathe a hypertonic saline solution from an ultrasonic nebulizer through a mouthpiece at saline concentrations of 3%, 4%, and 5%. After each inhalation period subjects be asked to cough up the expectorate in a sterile cup for analysis/quantitation of neutrophil cells influx
Nasal Epithelial Lavage Fluid (NELF) | measured (pre) before starting 6.6 hours of exposure, , immediately after (post), and at follow up 24 hours later (Follow Up)
  Saline is squirted into each nostril and filter paper is then inserted into each nostril for 2 minutes. NELF is then analyzed for acute phase proteins

CONTACTS AND LOCATIONS:
Locations (1):
- EPA Human Studies Facility, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No